CLINICAL TRIAL: NCT06474247
Title: Use of Postbiotic as Adjunct Treatment for Vaginal Candidiasis in Women
Brief Title: Postbiotic as Adjunct Treatment for Vaginal Candidiasis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Min-Tze LIONG (Other)
Collaborators: AIMST University (Unknown); Sumita Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Min-Tze LIONG, Professor, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIEC/INDT/APP/06/02/24-01
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Vaginal Candidiasis
Keywords: probiotic; postbiotic; vaginal candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postbiotic (Experimental): Postbiotic at 1g/day as an adjunct treatment against vaginal candidiasis in women for 4-weeks
  Interventions: Device: Postbiotic
- Placebo (Placebo Comparator): Placebo at 1g/day as an adjunct treatment against vaginal candidiasis in women for 4-weeks
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Postbiotic — Postbiotic at 1g/day as an adjunct treatment against vaginal candidiasis in women for 4-weeks
  Arms: Postbiotic
Device: Placebo — Placebo at 1g/day as an adjunct treatment against vaginal candidiasis in women for 4-weeks
  Arms: Placebo

SUMMARY:
This project aims to study the efficacy of intravaginal administration of postbiotic at 1g/day as an adjunct treatment against vaginal candidiasis in women for 4-weeks compared to placebo.

DETAILED DESCRIPTION:
Probiotics are live microorganisms that grant health effects to the host if consumed in sufficient amounts. Probiotic bacteria, which beneficially affect the host by improving the intestinal microbial balance, may affect the immune response, thus boosting the body system to combat against diseases. Meanwhile, postbiotic is an inactivated probiotic, probiotic-produced metabolites or their combination, which is capable of conferring beneficial effects to the host. Postbiotic has added advantages as compared to probiotic where inactivated cellular components remain potent though excluding any allergic factors, while the beneficial metabolites are applied directly to host upon administration and useful for applications such as skin topical use and intravaginal routes.

Vaginitis has been considered as one of the most common gynaecological conditions affecting women worldwide. Bacterial vaginosis and yeast vaginitis are two of three urogenital infections that affect as estimated one billion women in the world annually. The prevalence of vaginitis was reported to be varied from 5% to 50% among different study populations across major continents such as the United States of America, Europe and South Asia.

Vaginal candidiasis is one of the most common gynecological problems seen in primary care with Candida albicans account for 90% of the infection. The over-growth of this fungus in the vagina leads to a burning sensation in the vagina vulva, the production of heavy white/yellow curd-like discharge and/or an itchy vulva, puritus, dyspareunia, dysuria, irritation, soreness of the vulva and other discomforting symptoms that will ensure frequent hospital visits. The symptoms of vaginal candidiasis include vaginal itching or soreness, pain during sexual intercourse, pain or discomfort when urinating and abnormal vaginal discharge. Although most vaginal candidiasis is mild, some women can develop severe infections involving redness, swelling, and cracks in the wall of the vagina. It is also a most common form of fungal infection in pregnant mothers which may cause systemic infections in neonate particularly with low birth weight and prematurity after delivery.

Probiotics are preferred compared to antibacterial and antifungal drugs due to infection recurrence and drug resistance. It is a main concern that overuse of antibiotics could result in the development of antibiotic-resistant bacteria and fungus. Therefore, it is vital to find other alternatives to treat vaginal infections.

The maintenance of healthy vaginal microbiota is important for optimal vaginal microenvironment. Jang and team reported that intravaginal administration of probiotic mixture increased the regulation of vaginal IL-10 and Foxp3. As this may be due to the probiotic regulatory effects on immune responses in the vagina. A clinical study from Norway and Sweden found that the treatment with antibiotics or anti-fungal medication in combination with probiotics provided long-term cure against recurrence of vaginal candidiasis as compared to the control.

During the past several decades, the many published surveys of vaginal flora specimens obtained from asymptomatic women have clearly shown that C. albicans may be present without the typical symptoms of yeast vaginitis. In a study by Glover and Larsen, the results of successive cultures of vaginal flora specimens indicated that Candida species may be present in stable association with the genital epithelium. Moreover, the majority of women who have vaginal yeast also carry the organism in the gut.

In women, vaginal candidiasis has been related to emotional stress and suppression of immune system which step up the risk of Candida species overgrowth and become pathogenic. In addition, another study involving 512 women with candidiasiss reported a substantial negative impact on quality of life, with 42% feeling out of control of their lives and 60% feeling out of control of their bodies. Forty-one percent indicated a severe impact on their sexual lives. Meanwhile, 30% of women with recurrent episodes of candidiasis have reported considerable morbidity and suffering. The summary scores of the SF-36 in topic of subjective health status and health-related quality of life among women with Recurrent Vulvovaginal Candidosis (RVVC) in Europe and the USA also suggested that mental health was strongly affected by RVVC.

Current reports primarily emphasize on clinical effects of probiotics against candidiasis in women, with only few reports specifically on efficacy against recurrences. Very recent data are beginning to report on microbiota profiles of vaginal and feces of women with candidiasis, albeit rare. There have been no reports on these aspects from postbiotics. Information on proteins concentration, gene expression of vaginal microenvironment as affected by postbiotics against candidiasis are thus crucial. Thus, it is hoped that via this research, new scientific data is generated for future knowledge on these aspects, for use of postbiotics as an adjunct treatment against VC and RVVC.

ELIGIBILITY:
Inclusion criteria

* Women who are sexually active
* Confirmed with candidiasis as confirmed via clinical observations which include creamy whitish vaginal discharge and vulva-vaginal itchiness
* Willing to commit throughout the experiment

Exclusion criteria

* Long term medication (6 months or more) for any illnesses
* Pregnant
* Menopaused
* Uterus and/or cervix removed
* Cervical intraepithelial neoplasia
* Vaginal suppository treatments within 4-weeks prior to entering the study
* Oral medication for vaginal illnesses or any vaginal therapy such as hormones and estrogen within 4-weeks prior to entering the study
* Have used vaginal estrogen cream, ring or tablet within 4-weeks prior to entering the study
* Have used vaginal moisturizers, lubricants or homeopathic preparations within 4-weeks prior to entering the study
* Have used spermicide agent within 4-weeks prior to entering the study
* Have pelvic or any gynecologic surgery 6-months prior to entering the study

Ages: 18 Years to 81 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with vaginal candidiasis
Enrollment: 118 (Estimated)
Dates: Start 2024-06-02 (Actual); Primary Completion 2025-06-02 (Estimated); Study Completion 2025-06-02 (Estimated)

PRIMARY OUTCOMES:
Microbiota profiles of vaginal samples of women with vaginal candidiasis upon administration of postbiotic or placebo as assessed via next generation sequencing | 4-weeks
  Differences in microbiota abundance of vaginal samples of women with vaginal candidiasis upon administration of postbiotic compared to placebo

SECONDARY OUTCOMES:
Pathogenic yeasts profiles of vaginal samples of women with vaginal candidiasis upon administration of postbiotic or placebo as assessed via real time PCR | 4-weeks
  Differences in pathogenic yeasts abundance of vaginal samples of women with vaginal candidiasis upon administration of postbiotic compared to placebo
Quality of life profiles of women with vaginal candidiasis upon administration of postbiotic or placebo as assessed via questionnaires | 4-weeks
  Differences in quality of life parameters of women with vaginal candidiasis upon administration of postbiotic compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Sumita Bhatia, MD, Principal Investigator — Sumita Hospital
Locations (2):
- Sumita Hospital, Lucknow, Aliganj, India
- AIMST University, Bedong, Kedah, Malaysia

IPD SHARING:
Plan to Share IPD: No